CLINICAL TRIAL: NCT02165449
Title: Translational Biomarkers of Fast Acting Therapies in Major Depression
Brief Title: Biomarkers of Fast Acting Therapies in Major Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Narr, Associate Professor of Neurology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS001796; K24MH102743 (NIH); U01MH110008 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: ketamine; major depression; imaging; gene expression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Approved FDA indications for ketamine include use as an adjunct in the induction and maintenance of general anesthesia and for procedural sedation. For general anesthesia, ketamine is given at dosages ranging from 1-2mg/kg and given either as bolus injection or run continuously (0.1 to 0.3mg/kg/min) in conjunction with another anesthetic or sedation agent. In this study, ketamine at a subanesthetic dose of 0.5mg/kg will be diluted in 60cc of normal saline and administered via a slow IV infusion over 40 minutes at each treatment session in patients while undergoing hemodynamic monitoring. When used in this manner, ketamine infusion does not induce general anesthesia or states of unconsciousness, and patients remain fully awake, responsive to commands, and do not lose respiratory drive.

SUMMARY:
The drug Ketamine, available in medical practice since the late 1960s, is currently used for inducing general anesthesia or sedation during medical procedures. When given slowly as an injection into a vein, ketamine is shown to produce a very rapid effect on depression and to improve depressive symptoms within hours to days. By studying patients who receive a ketamine IV infusion, as an add-on treatment for depression, investigators may start to understand how changes in the brain or in gene function relate to getting better over a very short period of time. In this study, the investigators will enroll 60 patients currently ill with major depression selected to receive IV ketamine therapy under medical supervision. To study neurobiological changes relating to symptom improvement, the investigators will use advanced brain scans to measure brain structure, chemistry and function. Blood samples will measure changes in gene regulation and immune system response. Although some people have a rapid antidepressant response to ketamine, others do not respond. Also, antidepressant effects after ketamine usually wear off within days to weeks. We will determine if up to four doses of ketamine delivered two to three times a week may prolong antidepressant response to ketamine therapy. To determine the durability of ketamine treatment for depression, patients will be monitored by phone and via electronic devices twice a week for up to five weeks and will return for a final assessment when their symptoms return. For this trial, brain and blood sample measurements will occur before and after a patient receives their first ketamine infusion. Patients who do not remit after an initial dose of ketamine, will receive up to three additional ketamine treatments. Mood will be measured 24-hours after each subsequent ketamine infusion and brain and blood measurements be repeated at the time of remission or after the fourth ketamine infusion if remission does not occur. Patients will return for a final brain scan and blood sample when their depressive symptoms return or at five weeks if they continue remission. Investigators will able to see how changes brain measurements, gene regulation and immune response relate to improvements and relapse of depressive symptoms with ketamine IV therapy. The ketamine infusion sessions will occur at a special research unit (CTRC) at UCLA.

DETAILED DESCRIPTION:
Growing evidence implicates the glutamatergic system in the pathogenesis of depression, and receptor antagonists may provide a new generation of compounds for MDD treatment. In particular, the finding that the NMDA antagonist, ketamine, induces a rapid antidepressant response within hours to days has led to research investigating the neural mechanisms producing rapid antidepressant action and makes ketamine a valuable tool to identify biomarkers of depression response and of risk of relapse. The study of biomarkers for understanding the mechanistic actions of ketamine may serve to enhance emerging treatment approaches and provide new breakthroughs for translation of other drug targets.

Recently, the investigators of this trial have begun to offer off-label ketamine infusion treatment to clinical patients with treatment-resistant depression (TRD) and have developed a local treatment protocol for systematic clinical assessment, infusion monitoring and follow-up, which has been well-received and tolerated. The overarching goal of this study is to investigate imaging, gene expression and immune system biomarkers to help determine the underlying mechanisms and predictors for treatment response and relapse in MDD patients receiving ketamine and to compare these with the same biomarkers obtained from patients receiving ECT. The investigators aim to collect data from a sample of 60 patients who will receive serial infusions of ketamine, occurring 2-3 times a week, until they achieve remission or a total of 4 infusions. To study changes during or after ketamine treatment, we will use advanced brain scans that will allow us to measure brain structure, chemistry and function. We will also collect blood samples to measure changes in gene regulation and immune system response at the same time. Patients will also be assessed for basic cognitive function and mood. Brain and blood sample measurements will occur before ketamine infusion, 24 hours after the first infusion, after the 4th or last infusion, and at a final follow-up session approximately 5 weeks after ketamine treatment. We are also including remote mood assessment after treatment to more efficiently track relapse. We will therefore be able to see how changes over time in brain measurements and gene regulation, or immune response relate to improvements and relapse in depressive symptoms.

The investigators will address the following aims:

Aim 1: To use a comprehensive multimodal magnetic resonance imaging (MRI) battery including a) single voxel proton magnetic resonance spectroscopy (1HMRS), b) structural MRI (sMRI), c) arterial spin-labeling (ASL), d) resting state functional MRI (rs-fMRI) and e) diffusion MRI (dMRI) sensitive to different aspects of brain plasticity to isolate neurobiological markers linked with and predictive of ketamine response and subsequent relapse.

Hypothesis 1: Neuroplasticity in cortico-limbic (prefrontal and anterior cingulate cortex and hippocampus) and striatal networks, including changes in glutamate and other brain metabolites, in blood perfusion and in structural and functional connectivity will associate with therapeutic response to ketamine.

Aim 2: To use peripheral blood to measure inflammatory cytokines and their soluble receptors previously linked with depression or treatment outcome for the examination of relationships with ketamine response and subsequent relapse.

Hypothesis 2: Ketamine-induced symptom improvement will associate with altered concentrations of proinflammatory cytokines to indicate modulation of the immune response system.

Aim 3: To conduct transcriptome profiling using peripheral blood samples to identify gene expression correlates of ketamine response.

Hypothesis 3: Gene expression profiles will signal biological pathways underlying therapeutic response to ketamine.

Description of outcome measures:

1. Clinical outcome: The Hamilton Depression Rating Scale
2. Imaging markers: Image analysis will incorporate both standard and custom image analysis software and processing streams to measure changes neurochemistry, and structural and functional plasticity and connectivity occurring across time and in association clinical response. Specifically, outcome measures will include:

   1. Structural imaging and connectivity measures: combined volumetric and shape and diffusion metrics obtained from sMRI and dMRI data.
   2. Functional connectivity measures: Combined functional imaging measures obtained from resting state functional imaging data
   3. Neurochemistry: Brain metabolites including glutamate, choline, and NAA.
   4. Gene expression: Gene expression markers obtained from differential expression analyses.

Analyses: General linear mixed models and regression analyses will be used to determine changes across time and in association with clinical response for imaging markers. Weighted Gene Coexpression Network analysis (WGCNA) and Ingenuity Pathways analysis (IPA) will be used to identify functions and pathways associated with identified transcripts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 64 years, inclusive
* Diagnosis: DSM-IV TR criteria for non-psychotic major depression
* Hamilton Depression Rating Scale-17 item ≥ 18 or Montgomery Asberg Depression Scale ≥ 20
* A history of at least one previous major depressive episode prior to the current episode
* Recurrent Depression - in the current episode, have not responded to at least 2 adequate antidepressant trials (using Antidepressant Treatment History Form criteria)
* Have been continuously depressed for between 6-12 months
* Receiving approved monoaminergic antidepressant therapy
* No changes in antidepressant medication(s) in the past one (1) month
* Voluntary patient receiving ketamine
* Capacity to provide informed consent
* Have no contraindications to an adjunctive trial of ketamine infusion
* Be under the current care of a treating Psychiatrist
* If outpatient, a responsible driver available for transportation to and from scanning sessions
* Live locally, within travelling distance to UCLA
* Be available to participate for a 5-week research follow-up

Exclusion Criteria:

* Younger than 18 or older than 64
* Serious and imminent suicidal or homicidal risk (active suicidal ideations with or without a plan, HAM-D score ≥ 3 on item 3)
* Mental retardation or other developmental disorder
* Diagnosis of dementia of any type
* History of current substance abuse or dependence
* Psychotic reactions to medications, alcohol or illicit substances in the past
* Current or past history of psychosis, schizophrenia, bipolar disorder, delusional disorder or other psychotic disorder
* Treatment with medications with NMDA and NMDAR action
* Contraindication to ketamine
* Depression related to serious medical illness (i.e., mood disorder due to general medical condition)
* History of neurological disorder or other physical disorder (i.e. significant head injury) that could affect brain functioning
* Serious or unstable medical or neurological condition(s) that in the opinion of the treating physician or PI renders ketamine unsafe to administer
* Any condition that would contraindicate scanning (metal implants, claustrophobia or a breathing or movement disorder)
* Pregnancy (as confirmed by positive urine pregnancy test) or planning on becoming pregnant
* Non-English speaking (due to scales administered)
* Live outside of the Los Angeles area

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Rating Scale measured between baseline and 24 hrs following the first ketamine infusion treatment, and 24 hrs following up to three additional ketamine infusions | up to 2 weeks
  Change in mood ratings from the Hamilton Depression Rating Scale
Change in the Hamilton Depression Rating Scale measured between the last ketamine infusion treatment and 5 week follow-up | 5 weeks
  Change in mood ratings from the Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Change in gene expression measured between baseline and 24 hrs following the first ketamine infusion treatment, and 24 hrs following up to three additional ketamine infusions | up to 2 weeks
  Change in gene expression measured from peripheral blood
Change in gene expression measured between the last ketamine infusion treatment and 5 week follow-up | 5 weeks
  Change in gene expression measured from peripheral blood
Change in non-invasive Magnetic Resonance Imaging measures of structural connectivity measured between baseline and 24 hrs following the first ketamine infusion treatment, and 24 hrs following up to three additional ketamine infusions | up to 2 weeks
  Change in MRI measures of structural connectivity
Change in non-invasive Magnetic Resonance Imaging measures of structural connectivity measured between the last ketamine infusion treatment and at 5 weeks | 5 weeks
  Change in MRI measures of structural connectivity
Change in non-invasive Magnetic Resonance Imaging measures of functional connectivity measured between baseline and 24 hrs following the first ketamine infusion treatment, and 24 hrs following up to three additional ketamine infusions | up to 2 weeks
  Change in MRI measures of functional connectivity
Change in non-invasive Magnetic Resonance Imaging measures of functional connectivity measured between the last ketamine infusion treatment and at 5 weeks | 5 weeks
  Change in MRI measures of functional connectivity
Change in non-invasive Magnetic Resonance Imaging measures of neurochemistry measured between baseline and 24 hrs following the first ketamine infusion treatment, and 24 hrs following up to three additional ketamine infusions | up to 2 weeks
  Change in MRI measures of brain metabolite levels
Change in non-invasive Magnetic Resonance Imaging measures of neurochemistry measured between the last ketamine infusion treatment and at 5 weeks | 5 weeks
  Change in MRI measures of brain metabolite levels

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Narr, Ph.D., Principal Investigator — Geffen School of Medicine, University of California, Los Angeles (UCLA)
Locations (1):
- Geffen School of Medicine, UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data without protected health information will be shared according to approved UCLA IRB protocols.

REFERENCES:
- [Derived] Vasavada MM, Loureiro J, Kubicki A, Sahib A, Wade B, Hellemann G, Espinoza RT, Congdon E, Narr KL, Leaver AM. Effects of Serial Ketamine Infusions on Corticolimbic Functional Connectivity in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Jul;6(7):735-744. doi: 10.1016/j.bpsc.2020.06.015. Epub 2020 Jul 3. PMID 32900657
- [Derived] Sahib AK, Loureiro JRA, Vasavada MM, Kubicki A, Joshi SH, Wang K, Woods RP, Congdon E, Wang DJJ, Boucher ML, Espinoza R, Narr KL. Single and repeated ketamine treatment induces perfusion changes in sensory and limbic networks in major depressive disorder. Eur Neuropsychopharmacol. 2020 Apr;33:89-100. doi: 10.1016/j.euroneuro.2020.01.017. Epub 2020 Feb 12. PMID 32061453